CLINICAL TRIAL: NCT01452269
Title: Deaf Weight Wise: A Healthy Lifestyle Intervention for Deaf Adults
Brief Title: Study of a Healthy Lifestyle Intervention for Deaf Adults Who Are Overweight or Obese
Acronym: DWW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Steve Barnett, Director, Rochester Prevention Research Center, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Deaf Weight Wise
Record Dates: First submitted 2011-09-21; First posted 2011-10-14 (Estimated); Results first posted 2015-07-09 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate intervention group (Experimental): This arm will receive the intervention immediately following baseline data collection.
  Interventions: Behavioral: Deaf Weight Wise program
- Delayed intervention group (Experimental): This arm will receive the intervention one year following the immediate intervention group.
  Interventions: Behavioral: Deaf Weight Wise program

INTERVENTIONS:
Behavioral: Deaf Weight Wise program — Groups will consist of approximately 13 subjects who meet for 2 hours a week for 16 weeks. Group sessions will be offered at a variety of times and days of the week. A trained, deaf, ASL-fluent counselor will lead the sessions.
  Subjects will be asked to complete a food and physical activity diary. Each intervention session will include a weigh-in, group sharing/problem solving, discussion of a weight management topic, and goal setting/action planning for the next week. Periodically, each subject will receive a Personal Feedback Report. Subjects will be able to earn points for complying with various aspects of the program. Points can be redeemed for small prizes (i.e. water bottles).
  The maintenance phase consists of two meetings at the beginning of the 6-month maintenance period and three months later. This will consist of a weigh-in, review of self-monitored diet and physical activity, problem solving and goal setting/action planning for their long-term program.

SUMMARY:
The purpose of the Deaf Weight Wise study is to test a 16 week, evidence-based, comprehensive program to change obesity-related health behaviors in Deaf people who use American Sign Language (ASL) as their primary language.

Participants will be randomized to one of two study arms - immediate intervention or delayed intervention. In addition to the intervention activities, participants will also take part in five study visits over the course of two years. At these study visits, the investigators will administer several surveys as well as conduct biometric assessments.

The investigators primary hypothesis is that the immediate intervention group will increase their levels of physical activity and reduce their caloric intake and body weight immediately following the intervention, compared to the delayed intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Deaf men and women ages 40-70 years who use sign language and live in the Rochester Metropolitan Statistical Area (MSA), have a body mass index (BMI) of 25-45
* Permission to participate from a primary healthcare provider if: 1) self-reported diagnosis of a recent cardiovascular disease event (heart attack or stroke in past 6 months), and 2) self-reported heart condition, chest pain, dizziness, or other reason not to participate in physical activity 3) self-reported weight loss surgery in the past two years
* Must be willing to follow a healthy dietary pattern and to abstain from using weight loss medications during the study
* Must be willing and able to attend group sessions and to participate in data collection requirements

Exclusion Criteria:

* Participants who had a cardiovascular disease event in the past 6 months who did not obtain medical clearance from their provider
* Participants who had self-reported heart condition, chest pain, dizziness, or other reason not to participate in physical activity who did not obtain medical clearance from their provider
* Participants who had weight loss surgery in the past two years and who did not obtain medical clearance from their provider
* Pregnancy, breastfeeding, or planning a pregnancy during the study period (each of which will be determined by subject self-report through an in-person interview with a research team member)
* Those people who are unable or unwilling to provide written, informed consent
* Those people who are unable to see and interact with computer-based questionnaires and educational interventions

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2011-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Barnett, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester; National Center for Deaf Health Research, Rochester, New York, United States

REFERENCES:
- [Background] Samuel-Hodge CD, Johnston LF, Gizlice Z, Garcia BA, Lindsley SC, Bramble KP, Hardy TE, Ammerman AS, Poindexter PA, Will JC, Keyserling TC. Randomized trial of a behavioral weight loss intervention for low-income women: the Weight Wise Program. Obesity (Silver Spring). 2009 Oct;17(10):1891-9. doi: 10.1038/oby.2009.128. Epub 2009 Apr 30. PMID 19407810
- [Result] Barnett S, Matthews K, DeWindt L, Sutter E, Samuel-Hodge C, Yang H, Pearson TA; Deaf Weight Wise Study Group. Deaf Weight Wise: A novel randomized clinical trial with Deaf sign language users. Obesity (Silver Spring). 2023 Apr;31(4):965-976. doi: 10.1002/oby.23702. Epub 2023 Mar 8. PMID 36890106

RESULTS

PARTICIPANT FLOW:
Groups:
- Immediate Intervention Group: This arm received the Group intervention immediately following baseline data collection. Groups consisted of 4-12 subjects who meet for 2 hours a week for 16 weeks. Group sessions were offered at a variety of times. A trained, deaf, ASL-fluent counselor led the sessions.
  Subjects completed a food and physical activity diary. Each intervention session included a weigh-in, group sharing/problem solving, discussion of a weight management topic, and goal setting/action planning for the next week. Subjects received a Personal Feedback Report periodically. Subjects earned points for complying with various aspects of the program. Points were redeemed for small prizes (i.e. water bottles).
  The maintenance phase consisted of two meetings at the beginning of the 6-month maintenance period and three months later, and consisted of a weigh-in, review of self-monitored diet and physical activity, problem solving and goal setting/action planning for their long-term program.
- Delayed Intervention Group: This arm received the Group intervention one year following the immediate intervention group.Groups consisted of 4-12 subjects who meet for 2 hours a week for 16 weeks. Group sessions were offered at a variety of times. A trained, deaf, ASL-fluent counselor led the sessions.
  Subjects completed a food and physical activity diary. Each intervention session included a weigh-in, group sharing/problem solving, discussion of a weight management topic, and goal setting/action planning for the next week. Subjects received a Personal Feedback Report periodically. Subjects earned points for complying with various aspects of the program. Points were redeemed for small prizes (i.e. water bottles).
  The maintenance phase consisted of two meetings at the beginning of the 6-month maintenance period and three months later, and consisted of a weigh-in, review of self-monitored diet and physical activity, problem solving and goal setting/action planning for their long-term program.
Period: Overall Study
Arm/Group | Immediate Intervention Group | Delayed Intervention Group
Started | 48 | 56
Completed | 47 | 51
Not Completed | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Delayed Intervention Group: This arm received the intervention one year following the immediate intervention group.Groups consisted of 4-12 subjects who meet for 2 hours a week for 16 weeks. Group sessions were offered at a variety of times. A trained, deaf, ASL-fluent counselor led the sessions.
  Subjects completed a food and physical activity diary. Each intervention session included a weigh-in, group sharing/problem solving, discussion of a weight management topic, and goal setting/action planning for the next week. Subjects received a Personal Feedback Report periodically. Subjects earned points for complying with various aspects of the program. Points were redeemed for small prizes (i.e. water bottles).
  The maintenance phase consisted of two meetings at the beginning of the 6-month maintenance period and three months later, and consisted of a weigh-in, review of self-monitored diet and physical activity, problem solving and goal setting/action planning for their long-term program.
- Total: Total of all reporting groups
Arm/Group | Immediate Intervention Group | Delayed Intervention Group | Total
Number analyzed (Participants) | 48 | 56 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 53 | 97
  >=65 years | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (7.4) | 53.4 (7.8) | 53.5 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 39 | 71
  Male | 16 | 17 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 45 | 54 | 99
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 45 | 50 | 95
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 48 | 56 | 104
Became Deaf age 3 or younger [Number; unit: participants]
  Became Deaf age 3 or younger | 42 | 44 | 86
  Became Deaf age 4 or older, or unknown age | 6 | 12 | 18

OUTCOME MEASURES:

1. Primary Outcome: Weight Change
Description: We measured the mean change in weight for the immediate and delayed groups, from baseline to 6 months (post-intervention for the immediate group; no intervention yet for the delayed group). We used intention to treat analyses, with any missing values carried forward from baseline to the 6-month data point.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | Immediate Intervention Group | Delayed Intervention Group
Number analyzed (Participants) | 48 | 56
kilograms | -5.33 (0.88) | -1.98 (0.60)

2. Primary Outcome: Change in Dietary Risk Assessment (DRA) Score
Description: We measured the mean change in DRA score for the immediate and delayed groups, from baseline to 6 months (post-intervention for the immediate group; no intervention yet for the delayed group). We used intention to treat analyses, with any missing values carried forward from baseline to the 6-month data point. DRA scores range from 0-96; lower scores are better (improved dietary quality).
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: DRA score
Arm/Group | Immediate Intervention Group | Delayed Intervention Group
Number analyzed (Participants) | 48 | 56
DRA score | -6.3 (1.2) | -3.7 (1.3)

3. Primary Outcome: Change in Physical Activity Assessment (PAA) Score
Description: We measured the mean change in the moderate PAA score for the immediate and delayed groups, from baseline to 6 months (post-intervention for the immediate group; no intervention yet for the delayed group). We used intention to treat analyses, with any missing values carried forward from baseline to the 6-month data point. PAA moderate activity scores range from 0-27; higher scores are better (more physical activity).
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: moderate PAA score
Arm/Group | Immediate Intervention Group | Delayed Intervention Group
Number analyzed (Participants) | 48 | 56
moderate PAA score | 1.6 (0.5) | 1.0 (0.5)

ADVERSE EVENTS:
Time Frame: During the entire course of the study
Description: No adverse events occurred.
Arm/Group | Immediate Intervention Group | Delayed Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/56
Other Adverse Events (participants affected / at risk) | 0/48 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No